CLINICAL TRIAL: NCT03460743
Title: Evaluation of the Immunogenicity, Relative Efficacy, Safety and Reactogenicity of Flublok Quadrivalent® (Quadrivalent Recombinant Influenza Vaccine, Seasonal Formulation) Compared With a Marketed Quadrivalent Vaccine in Healthy Children and Adolescents Aged 3 to 17 Years-old.
Brief Title: Evaluation of a Recombinant Quadrivalent Influenza Vaccine Versus a Marketed Quadrivalent Inactivated Influenza Vaccine in Children 3 to 17.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Liomont (Industry)
Collaborators: EPIC Research CRO (Industry); ILS Clinical Research (Unknown); Q Square Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: LIO-04-16
Record Dates: First submitted 2018-03-04; First posted 2018-03-09 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Influenza, Human
Keywords: hemagglutinin influenza vaccine; recombinant influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Visit 1: screening visit, baseline blood sampling and administration of the study vaccine that can be performed on Day 0.
  Visit 1A and 2: Remote follow up contacts on day 2 and 7 post-vaccination. Visit 3: i. Follow up and blood sampling (for the 1-dose group); ii. Visit 3A, follow-up and application of the second dose of the vaccine (for the corresponding group); iii. Visit 3B, follow-up and blood sampling for the 2-dose group. The visits occur on Day 28.
  Months 3, 4, 5: Remote Contacts for safety tracking Visit 4: Remote contact for study closure and safety tracking at Month 6
Who Masked: Participant, Investigator
Masking Description: Participant- and observer-blind, the vaccine will be administered by a non-blinded vaccinator that will not participate in the clinical evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study group (Experimental): single or two doses of quadrivalent recombinant 180 ugm hemagglutinin influenza vaccine
  Interventions: Biological: Study group - quadrivalent recombinant hemagglutinin influenza vaccine
- Control group (Active Comparator): single or two doses of quadrivalent inactivated influenza vaccine.
  Interventions: Biological: Control group - quadrivalent inactivated influenza vaccine

INTERVENTIONS:
Biological: Study group - quadrivalent recombinant hemagglutinin influenza vaccine — Eligible subjects will be randomized, 1:1, to receive one or two doses of same vaccine. Subjects will be categorized in two age groups: subjects 9 to 17 years will be allocated in Group A and will receive one dose; Subjects 3 to 8 will be allocated to group B and the ACIP/CDC algorithm will be applied to determine should one or two doses will be applied 28 days apart. Vaccinator will be non blind and will not participate in the clinical evaluation.
  Arms: Study group
Biological: Control group - quadrivalent inactivated influenza vaccine — Eligible subjects will be randomized, 1:1, to receive one or two doses of same vaccine. Subjects will be categorized in two age groups: subjects 9 to 17 years will be allocated in Group A and will receive one dose; Subjects 3 to 8 will be allocated to group B and the ACIP/CDC algorithm will be applied to determine should one or two doses will be applied 28 days apart. Vaccinator will be non blind and will not participate in the clinical evaluation.
  Arms: Control group

SUMMARY:
Multicentric study, Phase III; this study is a randomized, participant- and observer-blind, parallel group evaluation to evaluate the immunogenicity, relative efficacy, safety and reactogenicity of a recombinant quadrivalent hemagglutinin influenza vaccine versus an inactivated quadrivalent influenza vaccine in pediatric subjects and adolescents of 3-17 years of age. Investigational vaccine is indicated for active immunization against influenza A and B for strains contained in the vaccine marketed in the United States for persons 18 years of age or older.

DETAILED DESCRIPTION:
Abbreviated title Evaluation of immunogenicity, relative efficacy, safety and reactogenicity of Flublok Quadrivalent® in healthy children and adolescents aged 3 to17 years.

Sponsor Product Identifiers Flublok® Quadrivalent of Laboratories Liomont, S.A. de C.V.

Flublok Quadrivalent consists of 180 μg total recombinant hemagglutinins Study Phase Phase 3 Study National multicentric Participating sites: Mexico: At least 10 research sites distributed in different states.

Clinical indication Vaccine indicated for active immunization against influenza A and B for strains contained in the vaccine; authorized in the United States for persons 18 years of age or older.

It will be evaluated in a population aged 3 to 17 years. Treatment Groups Flublok® Quadrivalent (research product) Fluzone® Quadrivalent (active comparator) Number of participants in the study 1,556 Estimated study duration: 25 months Duration of participation 6 months Randomization ratio 1:1 Study visits Visit 1: It corresponds to the screening visit, baseline blood sampling and administration of the study vaccine that can be performed on Day 0.

Visit 1A and 2: Remote contacts on day 2 and 7 post-vaccination. Visit 3: i. Follow up and blood sampling (for the 1-dose group); ii. Visit 3A, follow-up and application of the second dose of the vaccine (for the corresponding group); iii. Visit 3B, follow-up and blood sampling for the 2-dose group. The visits occur on Day 28.

Months 3, 4, 5: Remote Contacts for safety tracking Visit 4: Remote contact for study closure and safety tracking at Month 6. Statistical analysis plan • Primary efficacy analysis: Proportion of subjects in each age category and vaccine group who seroconvert, with seroconversion being defined as (a) a >4-fold rise in HAI antibody titer in those subjects seropositive (titer >10) at baseline or (b) achievement of an HAI titer of >40 in those seronegative at baseline. Seroconversion will be evaluated against each of the 4 vaccine antigens, on Study Day 28 (or Day 56 for 2-dose subjects), by category A and B separated

• Geometric Mean Titer (GMT) of HAI antibody against each vaccine antigen in each age category and vaccine group 28 days after immunization (Day 56 for 2-dose subjects) by category A and B separated Secondary efficacy analysis. Efficacy analysis and analysis of safety results associated to reactogenicity and other adverse events.

Final contribution of the study results The direct benefit for subjects, individually, is expected to be seasonal influenza protection with the expected degree of protection, specially among recipients of the IIV4 control vaccine, which is also approved for use in the age groups of the study population, evaluating in detail the comparative response of the research product.

The results of the study are intended to evaluate the immunogenicity, efficacy and safety of Flublok Quadrivalent in this population age and in this way, support the use of Flublok Quadrivalent for children and adolescents 3-17 years of age.

If the results are favorable and if the hypothesis is fulfilled, the extension of the indication to the evaluated age segment may result in greater protection of the child population so as, not to be unprotected by the limited resources in health, the shortage of vaccines in certain regions, and to improve the supply and accessibility of the population in general for influenza prevention.

The hypothesis underlying the study design and sample size estimated for the trial population from 3 to 17 years of age is based on the immunogenicity of Flublok Tetravalent, considering that the haemagglutination inhibition (HAI) seroconversion titers and the geometric mean of post-vaccination titers for the four hemagglutinin antigens in the vaccines after completion of vaccination with Flublok Quadrivalent are not inferior to those titers observed in those vaccinated with IIV4.

Statistical considerations. sample size is 330 subjects in each age cohort for each treatment group, reaching a power of 80% to detect a marginal difference of non-inferiority for the seroconversion rate between the groups of -0.1000. The seroconversion rate of the control group is 0.7000. The Flublok Quadrivalent seroconversion rate is assumed to be 0.6000 under the null hypothesis of inferiority. The power was estimated for the case that the relative seroconversion rate of Flublok Quadrivalent is 0.7000. The statistical test use is a one tailed Z test (unpooled). The significance level for the test was established in 0.0250.

A total of 1,556 subjects (330 complete cases per treatment group in subjects from 3 to 17 years of age) will be enrolled, considering possible losses up to a maximum of 15%.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 3 to 17 years.
* History of two previous influenza immunizations at any time, or influenza infection during the previous year.
* Female subjects of child-bearing potential (as defined by the onset of menses) must agree to prevent pregnancy and usage of an effective contraception, or having practiced sexual abstinence for at least 28 day prior to the first study vaccine administration. Female subjects of child-bearing potential must be tested for pregnancy within 24 hours prior to vaccine administration.
* In good general health, healthy or medically stable, as determined by the medical history, physical examination and the Investigator's judgment.
* Parent(s) or legal representative of each potential subject must comprehend the study requirements, sign the informed consent before any procedure, and agree to comply with planned study procedures and visits. Provide written consent prior to enrollment and initiation of any study procedure.
* Pediatric consent will be attained as per the Research Ethics Committee's determination when subject is aged 8 or older.

Exclusion Criteria:

* Known allergy to eggs (anaphylaxis, angioedema, respiratory distress), severe allergy (e.g. anaphylaxis) to other components of the vaccine or contraindications to receive the comparator IIV4.
* Use of systemic steroids at doses of 2mg/kg/day for more than 10 days of prednisone or its equivalent.

(The use of nasal or topical steroids will be allowed).

* Active neoplastic disease or a history of any malignancy.
* History of receiving the influenza vaccine within the previous 6 months.
* Plan to receive another influenza vaccine, during the study term.
* History of receiving immunoglobulin or another blood product within the 3 months prior to enrollment in this study.
* Acute or chronic medical condition that, in the opinion of the Investigator, would render immunization unsafe or would interfere with the evaluation of efficacy or the immune response to the vaccine.
* An acute illness, including a body temperature greater than 37.7°C, within 3 days prior to immunization.
* Receive an experimental vaccine or medication within 1 month prior to enrollment in this study, or the expectation to receive an experimental vaccine, medication, or blood product during the study period.
* Developmental delay, neurologic disorder, or seizure disorder requiring ongoing medical assistance (note: history of febrile seizure is not considered an exclusion criterion).
* History of Guillain-Barré syndrome within 6 weeks after the application a previous influenza vaccine.
* Concurrent participation in another clinical trial (active or follow-up phase).
* Any other condition or situation that would, in the opinion of the investigator, place them at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1556 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
Seroconversion | To be evaluated against each of the 4 vaccine antigens, on Day 28 (or Day 56 for 2-dose subjects), by category aged
  Proportion of subjects with seroconversion defined as (a) a >4-fold rise in HAI antibody titer in subjects seropositive (titer >10) at baseline or (b) an HAI titer of >40 in those seronegative at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Macias, MD, Study Chair — National Institute of Pediatrics
Locations (11):
- Mexico (11):
  - Clinical Research Institute Saltillo, Saltillo, Coahuila
  - Centro de Investigacion Clinica del Pacifico, Acapulco de Juárez, Guerrero
  - AMIC Pachuca, Pachuca, Hidalgo
  - Instituto Jalisciencie de Metabolismo, Guadalajara, Jalisco
  - AINPAD Morelia, Morelia, Michoacán
  - JM Research, Cuernavaca, Morelos
  - Instituto Nacional de Pediatria, Mexico City
  - CEMDEC, Mexico City
  - Clinical Research Institute Darwin, Mexico City
  - UDEP Puebla, Puebla City
  - Centro Especializado en Investigación Clínica CEIC, Veracruz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] King JC Jr, Cox MM, Reisinger K, Hedrick J, Graham I, Patriarca P. Evaluation of the safety, reactogenicity and immunogenicity of FluBlok trivalent recombinant baculovirus-expressed hemagglutinin influenza vaccine administered intramuscularly to healthy children aged 6-59 months. Vaccine. 2009 Nov 5;27(47):6589-94. doi: 10.1016/j.vaccine.2009.08.032. Epub 2009 Aug 27. PMID 19716456
- [Background] Baxter R, Patriarca PA, Ensor K, Izikson R, Goldenthal KL, Cox MM. Evaluation of the safety, reactogenicity and immunogenicity of FluBlok(R) trivalent recombinant baculovirus-expressed hemagglutinin influenza vaccine administered intramuscularly to healthy adults 50-64 years of age. Vaccine. 2011 Mar 9;29(12):2272-8. doi: 10.1016/j.vaccine.2011.01.039. Epub 2011 Jan 28. PMID 21277410